CLINICAL TRIAL: NCT04170868
Title: Psychoeducational Video Series - Proof of Concept
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 7850
Record Dates: First submitted 2019-11-12; First posted 2019-11-20 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Psychoeducation

STUDY DESIGN:
Intervention Model Description: The videos will be evaluated in a split-exposure clinical trial, whereby outpatients will be randomly assigned access to one of the two proof-of-concept videos for unlimited viewing. After ten days of access, the patients will spend an additional ten days without video access. The first ten-day procedure will then be repeated once over, with each participant now gaining access to the opposing proof-of-concept video. Clinical impairment data along with patient perspectives will be gathered at each transition junction for use in pre- and post-exposure analyses. The investigators hope to find meaningful improvements in patient functioning-along with a positive reception to the video format-such as to warrant further clinical investigation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Video 1 (Other): Ten-day exposure to one of two randomly assigned psychoeducational videos. Administration of outcome measures pre and post.
  Interventions: Other: ADHD Psycheducation
- Video 1 Washout (No Intervention): Ten-day washout period between access to the first and second videos.
- Video 2 (Other): Ten-day exposure to the second of the two randomly assigned psychoeducational videos. Administration of outcome measures pre and post.
  Interventions: Other: ADHD Psycheducation

INTERVENTIONS:
Other: ADHD Psycheducation — The videos will disseminate evidence-based strategies for the management of Attention Deficit Hyperactivity Disorder (ADHD). Each video, roughly two minutes, will both introduce the viewer to a single ADHD management strategy and explain how said strategy can effectively be integrated into their life.
  Arms: Video 1; Video 2

SUMMARY:
The purpose of this study is to produce and then assess a psychoeducational video series intended for use amongst an adult attention deficit/hyperactive clinical population. The videos will disseminate evidence-based strategies for the management of Attention Deficit Hyperactivity Disorder (ADHD). Each video, roughly two minutes, will both introduce the viewer to a single ADHD management strategy and explain how said strategy can effectively be applied. The collective of the finished video series will aim to cover the breadth of common ADHD-related issues. An example of the animated video styling can be found at the following link: bit.ly/ADHD_Ethics. The investigators will evaluate these videos in a proof of concept program, looking at outcomes in both functional skill development and patient perspective. The results will be presented in an undergraduate thesis presentation.

DETAILED DESCRIPTION:
The study will consist of four phases, each involving the completion of several self-report metrics following video exposure or the lack thereof. The investigators expect 30-40 patients to progress through a quadriphasic design.

Phase 1:

Upon understanding and signing an informed consent form, participants will complete a short demographics questionnaire that will enquire into their age, education level, and gender, but will not include specific identifying information such as name, initials, email, or home address.

Next, participants will be asked to complete a survey containing both the Tuckman Condensed Procrastination Scale (TCPS) and the Adult ADHD Self-Report Scale (ASRS). The data that are gathered from the ASRS will be used as a core inclusion-exclusion metric.

Finally, participants will be briefed on the video access system and then given their unique login credentials, which allow the investigators to track individual usage metrics. The investigators will then explain that for the next ten days the participant will have unlimited access to a single, randomly assigned experimental video (with participants split between one of two videos) adding that at the third and seventh days the participant will receive-pending consent-a friendly email reminder of their ability to access the video. Any questions will be addressed at this point.

All in, the time required to complete Phase 1 for a single participant will be 30-45 minutes.

Phase 2:

After ten days have elapsed, the participant will be sent an online survey link containing the TCPS, ASRS, and a Video Review Survey. The email will also explain how video access over the upcoming ten days will be restricted-as Phase 3 of the study commences-but that they need not worry as full-access will be reinstated following completion of the study. With that, participants will be reminded of the investigator's contact information and left to continue using the learned strategies for the upcoming ten days.

Phase 3:

Following the ten day washout period, participants will be sent another online survey link containing the TCPS and ASRS. The email will also contain access to the second of the two videos, along with a re-explanation of how the investigators hope they use it. From here, another ten-day exposure period will begin.

Phase 4:

After completing the second ten-day exposure period (totalling one month's time), the participant will be asked to answer a final Future Video Survey. Once the survey has been answered, the participant will have finished the study and will be thanked for their time. A contact address and number will be included in the email in the case of any unresolved question, and a link will be provided to reinstate participant video access.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and up
* Ability to fill out a computerized form
* Ability to access the Internet
* Ability/Willingness to watch several psychoeducational videos
* Ability/Willingness to understand and abide by the procedures and the acknowledge disclosure statement
* The participants in the ADHD group must be diagnosed by a psychiatrist. Diagnosis will be confirmed by re-evaluation using the Adult ADHD Self-Report Scale (ASRS)

Exclusion Criteria:

* Under 18 years of age
* Inability to fill out a computerized form
* Does not currently have Internet access
* Inability/Unwillingness to watch several psychoeducational videos
* Inability/Unwillingness to understand and abide by the procedures and acknowledge disclosure statement
* The participant has not been diagnosed with ADHD by a psychiatrist. Or, the diagnosis does not meet confirmation following re-evaluation using the Adult ADHD Self-Report Scale (ASRS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Tuckman Condensed Procrastination Scale (TCPS) Change (Video One) | Measured at days 0 and 10. Day 0 serves as a baseline for changes at Day 10 following exposure to video one.
  The TCPS is a 16-question condensed version of the original Tuckman Procrastination Scale and has been validated as the gold standard for the evaluation of procrastination proclivity. The TCPS assesses respondent behaviour by posing self-statements that can either be agreed or disagreed with on a four-point Likert-type scale. Out of the sixteen questions, five are reversed coded to promote accurate responding.
Tuckman Condensed Procrastination Scale (TCPS) Change (Video Two) | Measured at days 20 and 30. Day 20 serves as a quasi-baseline--following washout--for changes at Day 30 following exposure to video two.
  The TCPS is a 16-question condensed version of the original Tuckman Procrastination Scale and has been validated as the gold standard for the evaluation of procrastination proclivity. The TCPS assesses respondent behaviour by posing self-statements that can either be agreed or disagreed with on a four-point Likert-type scale. Out of the sixteen questions, five are reversed coded to promote accurate responding.

SECONDARY OUTCOMES:
Adult ADHD Self-Report Scale (ASRS) Change (Video One) | Measured at days 0 and 10. Day 0 serves as a baseline for changes at Day 10 following exposure to video one.
  The ASRS is an 18-item self-report screening scale used to assess adult ADHD. Each ASRS item contains a five-point scale where participants indicate how frequently they conduct themselves in the described manner; item responses can range from 'Never' to 'Very Often', where responses of 'Often' or 'Very Often' are consistent with ADHD typical dysfunction. When participant responses meet the criterion for ADHD typical dysfunction on at least 4 out of 6 screener items (denoted as 'Part A'), said participant will meet inclusion for the study. The remaining 12 ASRS items ('Part B') will be administered for use in the event that the screener criteria are met, and thus a need for further psychometric gradation arises.
Adult ADHD Self-Report Scale (ASRS) Change (Video Two) | Measured at days 20 and 30. Day 20 serves as a quasi-baseline--following washout--for changes at Day 30 following exposure to video two.
  The ASRS is an 18-item self-report screening scale used to assess adult ADHD. Each ASRS item contains a five-point scale where participants indicate how frequently they conduct themselves in the described manner; item responses can range from 'Never' to 'Very Often', where responses of 'Often' or 'Very Often' are consistent with ADHD typical dysfunction. When participant responses meet the criterion for ADHD typical dysfunction on at least 4 out of 6 screener items (denoted as 'Part A'), said participant will meet inclusion for the study. The remaining 12 ASRS items ('Part B') will be administered for use in the event that the screener criteria are met, and thus a need for further psychometric gradation arises.

OTHER OUTCOMES:
Video Review Survey (VRS) | Administered on day 10 and day 30. These are the points in which participants will have completed exposure to videos one and two, respectively.
  The VRS is a short questionnaire that participants will answer twice, each time following completion of a two-week video access block. The VRS requests participants to provide their opinions on the video-and the strategies contained within-that they had access to for the previous month. Through specific opinions, the investigators are better able to adapt future psychoeducational resources to the needs of people with ADHD.

IPD SHARING:
Plan to Share IPD: No
N/A as the data are a simple proof-of-concept.